CLINICAL TRIAL: NCT07097844
Title: A Comparison of the Efficacy of Sacral Erector Spinae Plane Block and Penile Block in Circumcision Surgery
Acronym: SACRAL ESP
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Siirt Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, ali kendal oğuz, specialist doctor in anestesiology and reanimation, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SAĞLIK BİLİMLERİ ÜNİVERSİTESİ
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Elective Circumcision Surgery
Keywords: Sacral ESPB; Penile Block; Pediatric Regional Anesthesia; Circumcision; FLACC Score; Opioid Consumption
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I - Sacral ESPB (Active Comparator): Type: Procedure
  Name: Sacral Erector Spinae Plane Block
  Description: Ultrasound-guided sacral ESPB using 0.8 mL/kg of 0.25% bupivacaine
  Interventions: Drug: 0.8 mL/kg of 0.25% bupivacaine
- Group II - Penile Block (Active Comparator): Type: Procedure
  Name: Penile Block
  penile block using 0.8 mL/kg of 0.25% bupivacaine
  Interventions: Drug: 0.8 mL/kg of 0.25% bupivacaine

INTERVENTIONS:
Drug: 0.8 mL/kg of 0.25% bupivacaine — 0.8 mL/kg of 0.25% bupivacaine

SUMMARY:
Effective perioperative analgesia is crucial for reducing hospital stay in pediatric surgical patients. Opioid-based analgesia, although effective, may lead to respiratory depression in the postoperative period. Therefore, alternative regional anesthesia techniques such as penile block and sacral ESPB are increasingly preferred.

Sacral ESPB provides both somatic and visceral analgesia by blocking the dorsal and ventral rami of the spinal nerves. It has the potential to block the pudendal nerve and achieve bilateral effect with a single midline injection. However, comparative data between sacral ESPB and penile block in circumcision surgeries is limited.

DETAILED DESCRIPTION:
Effective perioperative analgesia is crucial for reducing hospital stay in pediatric surgical patients. Opioid-based analgesia, although effective, may lead to respiratory depression in the postoperative period. Therefore, alternative regional anesthesia techniques such as penile block and sacral ESPB are increasingly preferred.

Sacral ESPB provides both somatic and visceral analgesia by blocking the dorsal and ventral rami of the spinal nerves. It has the potential to block the pudendal nerve and achieve bilateral effect with a single midline injection. However, comparative data between sacral ESPB and penile block in circumcision surgeries is limited.

In this prospective, double-blind, randomized controlled trial, 62 children aged 2 to 7 years undergoing elective circumcision at the Department of Pediatric Surgery of Diyarbakır Gazi Yaşargil Training and Research Hospital will be randomly assigned to two groups:

Group I will receive sacral ESPB using 0.8 mL/kg of 0.25% bupivacaine

Group II will receive a penile block using the same dosage and concentration.

Primary outcomes include intraoperative opioid use and postoperative rescue analgesic consumption within 24 hours. Secondary outcome includes time to discharge. Hemodynamic parameters and FLACC scores will be monitored at defined intervals.

ELIGIBILITY:
Inclusion Criteria:

ASA I pediatric patients aged 2-7 years

Scheduled for elective circumcision

Informed consent obtained from parents/legal guardians

Exclusion Criteria:

ASA score other than I

Age <2 or >7 years

Known allergy to local anesthetics

Refusal to participate

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
FLACC Pain Score | From arrival in the recovery room until 24 hours postoperatively
  Postoperative pain will be assessed using the FLACC (Face, Legs, Activity, Cry, Consolability) scale at 0, 15, 30, 45, 60, 90 minutes, and 2, 4, 6, 8, 10, 12, 18, and 24 hours after surgery. A FLACC score ≥4 will be treated with rescue analgesia.

SECONDARY OUTCOMES:
Total Perioperative Opioid and Rescue Analgesic Consumption | Up to 24 hours postoperatively
  Measured as total intraoperative fentanyl usage and postoperative administration of paracetamol and ibuprofen.

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing is currently under consideration. A final decision will be made after study completion and ethical approval.